CLINICAL TRIAL: NCT03562780
Title: Clinical Bioequivalence Study on Two Paracetamol Tablet Formulations
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Fortune Pharmacal Co., Ltd. (Industry)
Collaborators: Chinese University of Hong Kong (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: BABE-P18-107
Record Dates: First submitted 2018-06-08; First posted 2018-06-19 (Actual); Last update posted 2019-07-31 (Actual); Status verified 2019-06

CONDITIONS: Healthy
MeSH Terms: interventions — Acetaminophen

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fortolin Tab 500mg (Experimental): During the study session, healthy subjects will be administered a single oral dose of Fortolin Tab 500mg after an overnight fast of approximately 10 hours.
  Interventions: Drug: Fortolin Tab 500mg
- Panadol Caplet 500mg (Active Comparator): During the study session, healthy subjects will be administered a single oral dose of Panadol Caplet 500mg after an overnight fast of approximately 10 hours.
  Interventions: Drug: Panadol Caplet 500mg

INTERVENTIONS:
Drug: Fortolin Tab 500mg — Fortolin Tab 500mg is a generic product manufactured by Fortune Pharmacal Co. Ltd.
  Other Names: Acetaminophen Tablet 500mg
  Arms: Fortolin Tab 500mg
Drug: Panadol Caplet 500mg — Panadol Caplet 500mg is manufactured by GlaxoSmithKline (Dungarvan) Ltd.
  Other Names: Acetaminophen Caplet 500mg
  Arms: Panadol Caplet 500mg

SUMMARY:
The objective of the study is to compare the bioavailability of a generic product of paracetamol (immediate-release) with that of a reference product when administered to healthy volunteers under fasting condition. The test product is Fortolin Tab 500mg manufactured by Fortune Pharmacal Co. Ltd., and the reference product is Panadol Caplet 500mg manufactured by GlaxoSmithKline (Dungarvan) Ltd. The plasma pharmacokinetic data of paracetamol obtained from two formulations will be used to evaluate the interchangeability of the products.

ELIGIBILITY:
Inclusion Criteria:

1. Male and non-pregnant female, 18 to 55 years of age
2. Body Mass Index (BMI) between 18 to 25 kg/m2
3. Accessible vein for blood sampling
4. High probability for compliance and completion of the study
5. Female subjects who are surgically sterile or post-menopausal. Or female subjects of child bearing potential agree to practice abstinence or take effective contraceptive methods (e.g.implanted contraceptives, intra-uterine device or consistent condom plus spermicide use) from the start of screening until two weeks of last dose administration to prevent pregnancy.
6. Have signed the written informed consent to participate in the study.

Exclusion Criteria:

1. Clinically significant cardiovascular, hepatic, renal, gastrointestinal, neurological, psychiatric, metabolic and other diseases
2. Clinically significant abnormality in physical examination, vital signs, laboratory test results and ECG evaluation
3. Positive results of hepatitis B
4. Moderate smoker (more than 2 cigarettes a day within 3 months prior to the start of first dosing)
5. Moderate consumption of alcohol (more than one drink per day within 3 months prior to the start of first dosing)
6. Have lost or donated more than 350 ml of blood within 3 months prior to the start of first dosing
7. Subjects who are taking prescription or non-prescription medications (except for contraceptives, refer to "Inclusion Criteria" section) which is likely to be required during the course of the study
8. Use of paracetamol or other analgesic/antipyretic medications within 4 weeks before first dosing
9. Volunteer in any other clinical drug study within 2 months prior to the start of first dosing
10. Hypersensitivity to paracetamol or other drugs in its class
11. History of drug abuse in any form
12. Female subjects who are breastfeeding or pregnant
13. Subjects who are considered not suitable in participating the study due to other factors judged by investigators

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2018-11-30 (Actual); Primary Completion 2019-03-01 (Actual); Study Completion 2019-04-08 (Actual)

PRIMARY OUTCOMES:
Peak drug concentration (Cmax) of paracetamol | 12 hours
Area under the drug plasma concentration-time curve (AUC) of paracetamol | 12 hours

SECONDARY OUTCOMES:
Time to maximum concentration (Tmax) of paracetamol | 12 hours
Terminal elimination half-life (t1/2) of paracetamol | 12 hours

CONTACTS AND LOCATIONS:
Overall Officials: Prof. Zhong ZUO, Principal Investigator — School of Pharmacy, The Chinese University of Hong Kong; Dr. Andrea OY Luk, Study Director — Phase I Clinical Trial Centre, The Chinese University of Hong Kong
Locations (1):
- Phase 1 Clinical Trial Centre, The Chinese University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No